CLINICAL TRIAL: NCT01490450
Title: A Phase 2b, Randomized, Double-Blind, Placebo-Controlled, Dose Ranging, Multi-Center Study to Evaluate the Efficacy and Safety of BMS-945429 Subcutaneous Injection in Adults With Active Psoriatic Arthritis
Brief Title: Psoriatic Arthritis Dose Ranging Study for BMS-945429 in Subjects Who Are Not Responding to NSAIDs or Non-biologic Disease Modifying Anti-rheumatic Drugs (DMARDs) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM133-004; 2011-004016-29 (EudraCT Number)
Record Dates: First submitted 2011-11-14; First posted 2011-12-13 (Estimated); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — clazakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- PBO: Placebo matching BMS-945429 (Placebo Comparator)
  Interventions: Biological: Placebo matching BMS-945429
- BMS-945429 (25mg) (Experimental)
  Interventions: Biological: BMS-945429
- BMS-945429 (100mg) (Experimental)
  Interventions: Biological: BMS-945429
- BMS-945429 (200mg) (Experimental)
  Interventions: Biological: BMS-945429

INTERVENTIONS:
Biological: Placebo matching BMS-945429 — Injection, Subcutaneous, 0 mg, every 4 weeks, Short term:24 weeks, Long term: After 24 Wk, selected dose, open-label
  Arms: PBO: Placebo matching BMS-945429
Biological: BMS-945429 — Injection, Subcutaneous, 25 mg, every 4 weeks, Short term:24 weeks, Long term: After 24 Wk, selected dose, open-label
  Arms: BMS-945429 (25mg)
Biological: BMS-945429 — Injection, Subcutaneous, 100 mg, every 4 weeks, Short term:24 weeks, Long term: After 24 Wk, selected dose, open-label
  Arms: BMS-945429 (100mg)
Biological: BMS-945429 — Injection, Subcutaneous, 200 mg, every 4 weeks, Short term:24 weeks, Long term: After 24 Wk, selected dose, open-label
  Arms: BMS-945429 (200mg)

SUMMARY:
The purpose of this study is to characterize the safety, efficacy and dose response of BMS-945429 in subjects with active Psoriatic Arthritis and an inadequate response to Nonsteroidal anti-inflammatory drugs (NSAIDs) and non-biologic Disease modifying anti-rheumatic drugs (DMARDs).

ELIGIBILITY:
Inclusion Criteria:

* Must be on a stable background Methotrexate (MTX) therapy prior to Day1/Randomization. Subjects must have taken MTX for at least 3 months at a dose ≥ 15 mg/week to a maximum weekly dose of ≤ 25 mg/week, and be at a stable dose for 4 weeks prior to randomization (Day 1). Methotrexate dose ≥ 15 mg/week that was not efficacious and that was decreased due to toxicity as low as 10 mg/week is allowed
* Inadequate response to NSAID and/or non-biologic DMARD
* Minimum of 3 swollen and 3 tender joints
* Active psoriatic skin lesions over minimum 3% body surface area
* high sensitivity C-reactive protein (hsCRP) ≥ 0.3 mg/dL

Exclusion Criteria:

* Previously received or currently receiving concomitant biologic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (8):
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Denver Arthritis Clinic, Denver, Colorado
  - New England Research Associates, Llc, Trumbull, Connecticut
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Arthritis Associates Of Mississippi, Jackson, Mississippi
  - Box Arthritis And Rheumatology Of The Carolinas, Pllc, Charlotte, North Carolina
  - Health Research Of Oklahoma, Oklahoma City, Oklahoma
  - East Penn Rheumatology Associates, P.C., Bethlehem, Pennsylvania
- Argentina (2):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, San Miguel de Tucumán
- Australia (4):
  - Local Institution, Cairns, Queensland
  - Local Institution, Maroochydore, Queensland
  - Local Institution, Woodville, South Australia
  - Local Institution, Shenton Park, Western Australia
- Canada (4):
  - Manitoba Clinic, Winnipeg, Manitoba
  - Local Institution, Montreal, Quebec
  - Centre De Rhumatologie De L Est Du Quebec, Rimouski, Quebec
  - Centre De Recherche Musculo-Squelettique, Trois-Rivières, Quebec
- Czechia (2):
  - Local Institution, Pardubice
  - Local Institution, Prague
- Germany (3):
  - Local Institution, Bad Nauheim
  - Local Institution, Erlangen
  - Local Institution, Planegg
- Hungary (3):
  - Local Institution, Budapest
  - Local Institution, Debrecen
  - Local Institution, Veszprém
- Italy (2):
  - Local Institution, Florence
  - Local Institution, Napoli
- Mexico (3):
  - Local Institution, México, Aguascalientes
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Monterrey, Nuevo León
- Poland (5):
  - Local Institution, Bialystok
  - Local Institution, Dąbrówka
  - Local Institution, Elblag
  - Local Institution, Poznan
  - Local Institution, Warsaw
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Yaroslavl
- South Africa (4):
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Panorama, Cape Town, Western Cape
  - Local Institution, Pinelands, Cape Town, Western Cape
- Spain (3):
  - Local Institution, A Coruña
  - Local Institution, Barcelona
  - Local Institution, Seville

REFERENCES:
- [Derived] Mease PJ, Gottlieb AB, Berman A, Drescher E, Xing J, Wong R, Banerjee S. The Efficacy and Safety of Clazakizumab, an Anti-Interleukin-6 Monoclonal Antibody, in a Phase IIb Study of Adults With Active Psoriatic Arthritis. Arthritis Rheumatol. 2016 Sep;68(9):2163-73. doi: 10.1002/art.39700. PMID 27059799
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subcutaneous, every 4 weeks for 24 weeks
- Clazakizumab (25mg): Subcutaneous, 25 mg, every 4 weeks, for 24 weeks
- Clazakizumab (100mg): Subcutaneous, 100 mg, every 4 weeks, for 24 weeks
- Clazakizumab (200mg): Subcutaneous, 200 mg, every 4 weeks, for 24 weeks
Period: Period 1
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Started | 41 | 41 | 42 | 41
Completed | 38 | 40 | 38 | 33
Not Completed | 3 | 1 | 4 | 8
Not completed — Lack of Efficacy | 2 | 0 | 3 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 5
Not completed — Request to discontinue treatment | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 3
Not completed — No longer met study criteria | 0 | 1 | 1 | 0
Period: Period 2
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Started | 38 | 40 | 37 | 32
Completed | 36 | 39 | 37 | 28
Not Completed | 2 | 1 | 0 | 4
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg) | Total
Number analyzed (Participants) | 41 | 41 | 42 | 41 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 38 | 34 | 40 | 40 | 152
  >=65 years | 3 | 7 | 2 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (10.53) | 49.8 (14.05) | 49.3 (10.84) | 44.7 (13.75) | 47.9 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 20 | 20 | 86
  Male | 18 | 18 | 22 | 21 | 79

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Achieving American College of Rheumatology Criteria 20% Response Rate (ACR20)
Description: The ACR20/50/70 is a composite measure defined as both improvement of 20%, 50% or 70% in the number of tender and number of swollen joints, and a 20%, 50% or 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Time Frame: At 16 weeks
Population: Modified Intent-to-Treat (MITT) defined as all randomized subjects that received at least one dose of the study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 41 | 42 | 41
percentage of participants | 29.3 | 46.3 | 52.4 | 39.0

2. Secondary Outcome: Percent of Participants Achieving Psoriasis Area Severity Index (PASI) 75 Response Rate
Description: To calculate the PASI score, the psoriasis plaques found on each body region are graded for their combined redness, thickness, and scaliness. The severity of the plaques in each region is graded on a 0 to 4 scale, with 0 meaning no involvement and 4 meaning severe involvement. Next, the amount of surface area on each body region that is covered by the plaques is calculated. The total surface area affected by psoriasis is graded from 0 to 6, with 0 meaning no involvement and 6 meaning greater than 90 percent of the region covered in plaques.
  These grades are then fed into an equation to determine the patient's PASI score. The PASI score then is used as a clinical assessment of the patient's psoriasis involvement. A person free of psoriasis has a score of 0 and the score could be as high as 72.
  PASI 75 means that the person's PASI score dropped by 75 percent as a result of the psoriasis treatment.
Time Frame: Week 16 and Week 24
Population: MITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 41 | 42 | 41
percentage of participants
  week 16 | 14.6 | 12.2 | 16.7 | 4.9
  week 24 | 12.2 | 19.5 | 28.6 | 12.2

3. Secondary Outcome: Percent of Participants Achieving ACR50 and ACR70 Response Rate
Description: as for outcome 1
Time Frame: Week 16 and Week 24
Population: MITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 41 | 42 | 41
percentage of participants
  ACR50 (16 weeks) | 7.3 | 29.3 | 35.7 | 17.1
  ACR50 (24 weeks) | 14.6 | 34.1 | 35.7 | 24.4
  ACR70 (16 weeks) | 2.4 | 17.1 | 14.3 | 4.9
  ACR70 (24 weeks) | 4.9 | 19.5 | 23.8 | 12.2

4. Secondary Outcome: Percent of Participants Achieving ACR20 Response Rate at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: MITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 41 | 42 | 41
percentage of participants | 34.1 | 56.1 | 57.1 | 39.0

5. Secondary Outcome: Percent of Participants Achieving a Health Assessment Questionnaire (HAQ) Response
Description: For each item, there is a four-level difficulty scale that is scored from 0 to 3, representing normal (no difficulty) (0), some difficulty (1), much difficulty (2), and unable to do (3). There are 20 questions in eight categories of functioning - dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. The highest component score in each category determines the score for the category, unless aids or devices are required. Dependence on equipment or physical assistance increases a lower score to the level of 2 to more accurately represent underlying disability. The eight category scores are averaged into an overall HAQ score on a scale from zero (no disability) to three (completely disabled). The scale is not truly continuous but has 25 possible values (i.e., 0, 0.125, 0.250, 0.375 … 3).
  Response is measured by a reduction of at least 0.3 unit from baseline in HAQ index.
Time Frame: Weeks 16 and Week 24
Population: MITT
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 41 | 42 | 41
percentage of participants
  week 16 | 36.6 | 48.8 | 45.2 | 39.0
  week 24 | 26.8 | 51.2 | 47.6 | 36.6

6. Secondary Outcome: Mean Change From Baseline at Week 16 in Short Form (36) [SF-36] Scores
Description: The SF-36 questionnaire consists of eight scales yielding two summary measures: physical and mental health. The physical health measure includes four scales of physical functioning (10 items), role-physical (4 items), bodily pain (2 items), and general health (5 items). The mental health measure is composed of vitality (4 items), social functioning (2 items), role-emotional (3 items), and mental health (5 items). To score the SF-36, scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate better health status.
Time Frame: Baseline and Week 16
Population: MITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 40 | 40 | 41 | 39
score on a scale
  Mental component | 1.4 (1.507) | 1.2 (1.502) | 3.7 (1.478) | 1.1 (1.516)
  Physical component | 4.4 (1.236) | 6.5 (1.236) | 4.6 (1.217) | 4.1 (1.248)

7. Secondary Outcome: Mean Change From Baseline at Week 24 in SF-36 Scores
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: MITT
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 31 | 38 | 36 | 28
score on a scale
  Mental component | 3.6 (1.646) | 1.4 (1.538) | 3.9 (1.548) | 2.1 (1.689)
  Physical component | 4.9 (1.420) | 8.2 (1.360) | 5.7 (1.363) | 6.4 (1.461)

8. Secondary Outcome: Number of Participants With Anti-clazakizumab Antibodies
Time Frame: Up to 24 weeks
Population: MITT
Measure: Number; unit: participants
Arm/Group | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
Number analyzed (Participants) | 41 | 42 | 41
participants | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks per participant
Arm/Group | Placebo | Clazakizumab (25mg) | Clazakizumab (100mg) | Clazakizumab (200mg)
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 2/41 | 2/41 | 2/42 | 4/41
Other Adverse Events (participants affected / at risk) | 19/41 | 22/41 | 20/42 | 27/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Clazakizumab (25mg) (N=41) | Clazakizumab (100mg) (N=42) | Clazakizumab (200mg) (N=41)
Dystonia (Nervous system disorders) | 0 | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Adute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=41) | Clazakizumab (25mg) (N=41) | Clazakizumab (100mg) (N=42) | Clazakizumab (200mg) (N=41)
Nasopharyngitis (Infections and infestations) | 1 | 6 | 2 | 4
Pharyngitis (Infections and infestations) | 4 | 4 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 6 | 0 | 3 | 1
Urinary tract infection (Infections and infestations) | 2 | 4 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 9 | 6 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 6 | 4 | 4
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 1 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 5 | 2 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Gastritis (Gastrointestinal disorders) | 1 | 4 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1
Injection site reaction (General disorders) | 1 | 4 | 1 | 2
Injection site erythema (General disorders) | 0 | 0 | 3 | 3
Headache (Nervous system disorders) | 4 | 3 | 2 | 1
Migraine (Nervous system disorders) | 3 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No